CLINICAL TRIAL: NCT01596816
Title: Intermediate-risk Prostate Cancer : Assessment of Hypofractionated Stereotactic Boost - Prospective Phase II Study
Brief Title: Hypofractionated Stereotactic Boost in Prostate Cancer
Acronym: CKNO-PRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKNO-PRO-0901; 2010-A00237-32 (Other: IDRCB Number (ANSM_DEDIM))
Record Dates: First submitted 2011-06-15; First posted 2012-05-11 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Boost by CyberKnife (Experimental)
  Interventions: Radiation: First part of treatment : Conformal irradiation; Procedure: Fiducials placement; Radiation: Second part : hypofractionated stereotactic boost
- Boost by linear accelerator (Experimental)
  Interventions: Radiation: First part of treatment : Conformal irradiation; Procedure: Fiducials placement; Radiation: Second part : hypofractionated stereotactic boost

INTERVENTIONS:
Radiation: First part of treatment : Conformal irradiation — 23 fractions (2 Gy/session), are delivered over 42 days maximum, for a total dose of 46 Gy
Procedure: Fiducials placement — Placement of intra-prostatic markers for the tracking
Radiation: Second part : hypofractionated stereotactic boost — 3 fractions (6Gy/session) are delivered over 5 to 9 days (at least 48 hours between sessions) for a total dose of 18 Gy

SUMMARY:
hypofractionated stereotactic boost radiation (prostate) after normofractionated radiotherapy (prostate + seminal vesicles).

DETAILED DESCRIPTION:
The aim of this study is to assess the safety of hypofractionated stereotactic boost radiation (prostate) after normofractionated radiotherapy (prostate + seminal vesicles).

ELIGIBILITY:
Inclusion Criteria:

* Prostate adenocarcinoma proved by histology
* With at least one of this intermediate-risk criterias:

  * T2b
  * and/or PSA between 10 et 20 ng/ml
  * and/or Gleason score = 7
* Prostatic volume ≤ 80 cc
* No adenopathy(lymph node < 1.5 cm on scanner or MRI and/or in lymph node dissection)
* No metastasis (bone scan)
* Age >= 18 ans
* No prior pelvic irradiation
* No prior anticancer treatment (prostatectomy, chemotherapy, hormonotherapy > 3 months)
* Performance status (ECOG) < 1
* No contraindication of fiducials implantation, hemostasis disorders must be treated before the implantation
* Life expectancy >= 10 weeks
* Patient affiliated to health insurance
* Informed consent signed by the patient

Exclusion Criteria:

* Cancer no histologically proved
* Unfavorable-risk(T2c and/or PSA > 20 ng/ml and/or Gleason > 7)
* Favorable-risk(T1c T2a and PSA < 10 ng/ml and Gleason < 7)
* T3 and T4
* History of cancer uncontrolled and/or treated since less of 5 years (except basal cell carcinoma of the skin)
* Contraindication to MRI
* IPSS score > 10
* Recurrent or metastatic disease
* Allergy to gold
* Patient already included in another therapeutic trial with an experimental molecule
* Unable for medical follow-up (geographic, social or mental reasons)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in rectal functions | Every 3 months after boost irradiation during 1 year and then every 6 months during 2 years
  * Assessment of rectal toxicity according to the NCI-CTCAE v4.0 scale.
  * Acute toxicities are defined as all toxicities occurring within 6 months after the start of radiotherapy, late toxicities are those that occur beyond this period.
Change from baseline in urinary function. | Every 3 months after boost irradiation during 1 year and then every 6 months during 2 years
  * Assessment of urinary toxicity according to the NCI-CTCAE v4.0 scale.
  * Acute toxicities are defined as all toxicities occurring within 6 months after the start of radiotherapy, late toxicities are those that occur beyond this period.

SECONDARY OUTCOMES:
Local control of prostate cancer | 3 years
  Local control is defined as:
  * Non progressive PSA according to Phoenix criteria
  * Non progressive clinical examination (DRE)
  * No pathological findings on MRI
Global and metastase-free survival | Up to 5 years after treatment
  Time measurement between the inclusion and the date of death/metastatic progression
PSA kinetics | Between radiotherapy and boost, and after treatment : every 3 months
  Comparison of the PSA dosage before, at the end of treatment then every 3 months. The PSA dosage evolution will be correlate with the local control treatment.
Sexual toxicity | Up to 5 years after treatment
  According to IIEF5 questionnaire ( International Index of Erectile Function )
Technical criteria : Fiducial placement (yes/no) | During the time of treatment
Urinary discomfort | Up to 5 years after treatment
  According to IPSS questionnaire ( International Prostate Symptom Score)
Technical criteria : Cumulative dosimetry (1 time/ 2 times) | During the time of treatment
Technical criteria : boost schedule (yes/no) | During the time of treatment
Technical criteria : duration of boost | During the treatment
  Time between patient's entry and exit of the radiotherapy treatment room

CONTACTS AND LOCATIONS:
Overall Officials: Eric LARTIGAU, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (7):
- France (7):
  - Centre Paul Papin, Angers
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar LAMBRET, Lille
  - Centre Léon Bérard, Lyon
  - Val d'Aurelle-Paul Lamarque, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquier D, Nickers P, Peiffert D, Maingon P, Pommier P, Lacornerie T, Martinage G, Tresch E, Lartigau E. Hypofractionated stereotactic boost in intermediate risk prostate carcinoma: Preliminary results of a multicenter phase II trial (CKNO-PRO). PLoS One. 2017 Nov 30;12(11):e0187794. doi: 10.1371/journal.pone.0187794. eCollection 2017. PMID 29190707